CLINICAL TRIAL: NCT05080257
Title: Prognostic Value Of Chest Ultrasound (Lung Ultrasound Score) In COVID-19 Pneumonia Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karim Osama Mohammed Sleem, Resident, Chest Department, Principal investigator, Medical Doctor, Assiut University
Other Study IDs: Prognostic value of LUS COVID
Record Dates: First submitted 2021-10-06; First posted 2021-10-15 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Lung Ultrasonography — The ultrasonography will be done using the curved probe of the SONOACE R3 SAMSUNG ultrasonography machine, SN: S0GYM3HCC00016M, manufacture date: 12-2012.
  Assessment of lung condition using the Lung Ultrasonography Score (total score calculated from the 12 standard examined areas, from 0 to 3 in each area, with a minimum of 0 up to 36)

SUMMARY:
This study aims to

1. To study the prognostic value of LUS in COVID-19 patients.
2. To assess the relation between Lung Ultrasonography Score and disease severity in COVID-19 Patients.
3. To assess the relation between Lung Ultrasonography Score and mortality in COVID-19 patients.

DETAILED DESCRIPTION:
At the end of 2019, the COVID-19 pandemic broke out in Wuhan, China, and within few months -in March 2020- it was declared a pandemic by the WHO.

As of September 15th ,2021, there have been 226,844,344 confirmed cases of COVID-19, including 4,666,334 deaths, reported to WHO (1).

Due to the prevalence of COVID-19 and the financial burden it puts on the healthcare system, the use of a simple, affordable and reliable imaging modality was necessary.

The main idea in this research will be evaluating the value of Lung Ultrasonography Score in predicting the prognosis of patients with COVID-19 pneumonia and investigate the presence of a relation between the Lung Ultrasonography Score and patients' prognosis and mortality (2).

* Currently, Lung ultrasound had sensitivity 86%, specificity 71.6%, NPV 81.7%, and PPV 77.7%. The LUS had an area under the curve of 0.84 (95% CI 0.78, 0.90). When including examinations visualizing twelve lung areas, lung US had sensitivity 90.9% and specificity 75.6%, with NPV 87.2% and PPV 82.0% and an area under the curve of 0.89 (95% CI 0.83, 0.96). (3).
* In COVID-19 patients admitted in ED, LUS was a good predictor of death, ICU admission, and endotracheal intubation.
* Our main strategy will be enrolling patients admitted to the chest department's isolation unit, conduct clinical examination, laboratory investigations and imaging and conduct chest ultrasonography and calculate the Lung Ultrasonography Score of the patients and create a correlation between the Lung Ultrasonography score and their prognosis and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18.
* All Confirmed COVID-19 Patients by PCR or highly suspected patients admitted to the chest department's isolation unit during the duration of the study.

Exclusion Criteria:

* Age < 18.
* Heart Failure
* Chronic lung diseases with similar ultrasonographic findings to COVID-19 (ILD, Bronchiectasis, old T.B).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample size calculation will be carried out using G*Power 3 software , A minimum calculated sample of 60 COVID-19 cases will be needed to detect an effect size of 0.2 (22%-70%) vs (40%-93%) in the diagnostic yield (sensitivity and specificity) of lung US in severity of COVID-19 diagnosis, with an error probability of 0.05 and 80% power on a one-tailed test
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between Lung Ultrasonography Score and condition severity (inflammatory markers) | through study completion, an average of 2 years.
  creation of a statistical relation between the Lung Ultrasonography Score and the severity of the condition, which is assessed by clinical examination and inflammatory markers.
Mortality | Through study completion, an average of 2 years.
  creation of a statistical relation between the Lung Ultrasonography Score and mortality.

SECONDARY OUTCOMES:
Ventilatory support. | Through study completion, an average of 2 years.
  creation of a statistical relation between the Lung Ultrasonography Score and the ventilatory support needed by the patients.
Duration of hospital stay | Through study completion, an average of 2 years.
  Assessment of relation between Lung Ultrasonography Score and the duration of hospital stay.
ICU Admission | Through study completion, an average of 2 years.
  Assessment of relation between Lung Ultrasonography Score and the ICU admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: WHO dashboard for updated COVID-19 statistics — http://covid19.who.int/
- See also: 2- Proposal for International Standardization of the Use of Lung Ultrasound for Patients With COVID-19, Journal of Ultrasound in Medicine, volume 39 issue 7 — http://onlinelibrary.wiley.com/doi/full/10.1002/jum.15285
- See also: 3- Brenner, D.S., Liu, G.Y., Omron, R. et al. Diagnostic accuracy of lung ultrasound for SARS-CoV-2: a retrospective cohort study. Ultrasound J 13, 12 (2021) — https://theultrasoundjournal.springeropen.com/articles/10.1186/s13089-021-00217-7
- See also: 4- Faul, F., Erdfelder, E., Lang, A.-G. & Buchner, A. (2007). G*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behavior Research Methods, 39, 175-191 — https://link.springer.com/article/10.3758/BF03193146
- See also: 5- de Alencar, J.C.G., Marchini, J.F.M., Marino, L.O. et al. Lung ultrasound score predicts outcomes in COVID-19 patients admitted to the emergency department. Ann. Intensive Care 11, 6 (2021). https://doi.org/10.1186/s13613-020-00799-w — https://annalsofintensivecare.springeropen.com/articles/10.1186/s13613-020-00799-w